CLINICAL TRIAL: NCT03315832
Title: Efficacy of Angiotensin Receptor Blocker Following aortIc Valve Intervention for Aortic STenOsis: a Randomized mulTi-cEntric Double-blind Phase II Study
Acronym: ARISTOTE
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: problem of faisability
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: I16007 (ARISTOTE)
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Aortic Valve Stenosis; Valsartan; Angiotensin Receptor Antagonists; Transcatheter Aortic Valve Replacement; Heart Valve Prosthesis Implantation; Hypertrophy, Left Ventricular
Keywords: Aortic Valve Stenosis; Valsartan; Angiotensin Receptor Antagonists; Transcatheter Aortic Valve Replacement; Heart Valve Prosthesis Implantation; double-blind phase II study; left ventricular mass
MeSH Terms: conditions — Aortic Valve Stenosis; Hypertrophy, Left Ventricular | interventions — Valsartan

STUDY DESIGN:
Intervention Model Description: Patients with the diagnosis of severe AS and indication for valve intervention (i.e. SAVR or TAVR) fulfilling all inclusion/exclusion criteria will be randomized using 1:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Valsartan (Experimental): The active treatment is valsartan, an orally active, potent, and specific angiotensin II receptor antagonist. The treatment will be initiated (80 mg, daily) at 5±4 days following aortic valve intervention. The dose will be increased at 160 mg daily 13±2 days after aortic valve intervention and, if well tolerated, for the remaining period of the study.
  Interventions: Drug: Valsartan
- Placebo Oral Tablet (Placebo Comparator): The comparative treatment will be a placebo; tablets of valsartan and placebo have a similar appearance and administration mode. Patient in the control group will receive a placebo using the same protocol as the valsartan group.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Valsartan — The active treatment is valsartan, an orally active, potent, and specific angiotensin II receptor antagonist. The treatment will be initiated (80 mg, daily) at 5±4 days following aortic valve intervention. The dose will be increased at 160 mg daily 13±2 days after aortic valve intervention and, if well tolerated, for the remaining period of the study.
  Arms: Valsartan
Drug: Placebo Oral Tablet — The comparative treatment will be a placebo; tablets of valsartan and placebo have a similar appearance and administration mode. Patient in the control group will receive a placebo using the same protocol as the valsartan group.
  Arms: Placebo Oral Tablet

SUMMARY:
Aortic stenosis (AS) is the most frequent valvular heart disease in Western countries, with increasing prevalence. Recent guidelines recommend aortic valve intervention (surgical aortic valve replacement [SAVR] or transcatheter aortic valve replacement [TAVR]) in severe AS, as soon as symptoms or left ventricular (LV) dysfunction occur, in order to improve clinical outcome and achieve LV mass (LVM) regression. The highest amount of LVM regression is obtained during the first year. Nevertheless, there is heterogeneity in LV remodeling and residual LV hypertrophy is associated with poorer postoperative improvement in cardiac function and morphology. Incomplete regression of LV hypertrophy at 12 months after SAVR is a powerful predictor of adverse outcome. Yet, the use of specific pharmacological therapy to improve postoperative LVM regression could be an appealing therapeutic option after aortic valve intervention.

Renin-angiotensin-aldosterone system blockers (RAASb) and more particularly angiotensin-II receptor blockers (ARBs) are efficient in reducing LVM in hypertensive patients, as emphasized by several meta-analyses. In addition, ARBs improve myocardial relaxation, diastolic function, decreased hypertrophy and may have anti-fibrotic effects. In a recent retrospective study from our group, RAASb prescription after SAVR was associated with increased survival, but confirmation through a randomized trial is mandatory. In a prospective randomized single-center study, the use of candesartan was associated both with LV and LA remodeling as compared to the conventional management. Nevertheless, these results are based on echocardiographic data, which is not the gold standard for the assessment cardiac remodeling, and no placebo or active comparator was tested to control the impact of ARBs in these patients.

The primary objective of this Phase II study is to investigate the efficacy of valsartan, introduced postoperatively, as compared to placebo, on 1-year changes in indexed LVM, as assessed by CMR, in patients undergoing aortic valve intervention (SAVR or TAVR) for AS.

The secondary objectives are to compare the efficacy of valsartan vs. placebo in terms of one-year changes (difference from baseline) in cardiac function and in cardiac morphology, one-year exercise capacity and one-year changes in biomarkers related to cardiac function. In addition, the assessment of the safety of valsartan will also be considered as secondary objective.

The ARISTOTE trial is a multicenter prospective phase II, randomized, double-blind study including patients with the diagnosis of severe AS and indication for valve intervention.

The active treatment is valsartan, an orally active, potent, and specific angiotensin II receptor antagonist.

Patients will be randomized between 2 groups (valsartan versus placebo) and the treatment will be initiated (80 mg daily) at 5±4 days following aortic valve intervention. The comparative treatment will be a placebo; tablets of valsartan and placebo have a similar appearance and administration mode. Patient in the control group will receive a placebo using the same protocol as the valsartan group.

The patients will be cautiously monitored and any adverse events will be collected. The dose will be increased at 160 mg daily 13±2 days after aortic valve intervention and, if well tolerated, for the remaining period of the study. The tolerance will be regularly assessed and dose adjusted according to a pre-specified algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Men with age ≥18 years
* Women at postmenopausal state as defined by absence of menses for the last 12 months without alternative medical cause.
* Severe AS, defined according most recent guidelines (aortic valve area <1.0cm² or <0.6cm²/m² and aortic mean pressure gradient ≥40mmHg or aortic maximal velocity >4m/s, as assessed using transthoracic echocardiography [TTE]).
* Indication for aortic valve intervention
* Affiliation to the French Social Security system
* Signed informed consent.

Exclusion Criteria:

* Patients already under any Renin-Angiotensin-Aldosterone System blockers (RAASb) prior to randomization.
* Concomitant coronary artery bypass graft or other valvular intervention
* Other significant left-sided valvular heart diseases (≥moderate), even without concomitant procedure
* Any contra-indication to CMR
* Chronic kidney disease with estimated glomerular filtration rate (GFR) <30 ml/min
* Prior or planned organ transplantation
* Hyperkaliemia (kaliemia >5.5 mmol/L at inclusion visit)
* Severe hepatic failure, biliary cirrhosis, cholestasis
* Combined use of aliskiren and concomitant diabetes mellitus or renal failure with GFR<60mL/min/1.73m²
* Low systolic blood pressure (<100mmHg)
* History of angioedema
* History of hypersensitivity or allergy to Angiotensin-II Receptor Blockers or excipient
* Under legal authority.
* Unwilling to consent

Secondary Exclusion Criteria:

* Patients not under RAASb prior to randomization but who should benefit from this treatment to improve outcome:
* Heart failure with reduced ejection fraction (<40%)
* Coronary artery disease
* Clinical peripheral artery disease
* History of cerebrovascular disease
* Uncontrolled hypertension despite the use of other therapeutic classes
* Diabetes mellitus
* Impossibility to perform randomization into the 9-day post-intervention period due to per procedural complication with prolonged stay in intensive cardiac care unit (including death).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-02 (Estimated); Primary Completion 2025-07-02 (Estimated); Study Completion 2025-07-02 (Estimated)

PRIMARY OUTCOMES:
Indexed left ventricular mass | Day 0 to Year 1
  the 1-year change from baseline in indexed LVM after aortic valve intervention as assessed using cardiac magnetic resonance (CMR)

SECONDARY OUTCOMES:
Left ventricular global longitudinal strain | Day 0 to Year 1
  The 1-year change from baseline in left ventricular global longitudinal strain quantified using CMR
Left ventricular global longitudinal strain | Day 0 to Year 1
  The 1-year change from baseline in Left ventricular global longitudinal strain quantified using transthoracic echocardiography (TTE)
Left atrial volume | Day 0 to Year 1
  The 1-year change from baseline in Left atrial volume quantified using CMR
Left atrial volume | Day 0 to Year 1
  The 1-year change from baseline in Left atrial volume quantified using TTE
Indexed left ventricular mass | Day 0 to Year 1
  the 1-year change from baseline in indexed LVM after aortic valve intervention as assessed using TTE (real-time 3D)
Native T1 | Day 0 to Year 1
  the 1-year change from baseline in native T1 using CMR
Rate of late gadolinium enhancement (LGE) | Day 0 to Year 1
  the 1-year change from baseline in rate of LGE using CMR
Volume of late gadolinium enhancement (LGE) | Day 0 to Year 1
  the 1-year change from baseline in volume of LGE using CMR
Extra cellular volume | Day 0 to Year 1
  The 1-year change from baseline in extra cellular volume using CMR
Indexed interstitial volume | Day 0 to Year 1
  The 1-year change from baseline in Indexed interstitial volume using CMR
Electrocardiographic strain | Day 0 to Year 1
  The 1-year change from baseline in Electrocardiographic strain
Left ventricular ejection fraction | Day 0 to Year 1
  The 1-year change from baseline in Left ventricular ejection fraction using CMR
Left ventricular ejection fraction | Day 0 to Year 1
  The 1-year change from baseline in Left ventricular ejection fraction using TTE
Peak exercise VO2 | Year 1
  The 1-year measurement of Peak exercise VO2
VE/VCO2 ratio | 1 year
  The 1-year measurement of VE/VCO2 ratio
Maximal load | 1 year
  The 1-year maximal load reached
New-York heart association functional class | 1 year
  The 1-year assessment of New-York heart association functional class
Exercise oscillatory ventilation rate | 1 year
  The 1-year quantification of exercise oscillatory ventilation rate
Nt-pro Brain natriuretic peptide | Day 0 to Year 1
  The 1-year change from baseline in level of Nt-pro Brain natriuretic peptide using immunoassay
Plasma cardiac troponin I | Day 0 to Year 1
  The 1-year change from baseline in concentration of Plasma cardiac troponin I using high-sensitivity assay
Incidence of treatment-Emergent Adverse Events | Day 1 to Month 13
  Clinical occurrence of adverse events (AEs) and serious adverse events (SAEs) during the duration of the study period ending month 13

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges university hospital, Limoges, France